CLINICAL TRIAL: NCT01210807
Title: Clinical Evaluation of the One-Piece Tecnis Multifocal IOL, Model ZMB00
Brief Title: Clinical Evaluation of the One-Piece Tecnis Multifocal Intraocular Lens (IOL)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DIOL-105-TMF1
Record Dates: First submitted 2010-06-17; First posted 2010-09-29 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multifocal Intraocular Lens (Experimental): ZMB00 multifocal intraocular lens
  Interventions: Device: One-Piece Tecnis Multifocal IOL
- Monofocal Intraocular Lens (Active Comparator): ZCB00 monofocal intraocular lens
  Interventions: Device: One-Piece Tecnis monofocal IOL, Model ZCB00

INTERVENTIONS:
Device: One-Piece Tecnis Multifocal IOL — One-piece Tecnis Multifocal IOL, Model ZMB00, implanted lens.
  Other Names: Model ZMB00
  Arms: Multifocal Intraocular Lens
Device: One-Piece Tecnis monofocal IOL, Model ZCB00 — Control lens: One-Piece Tecnis monofocal IOL, Model, ZCB00, implanted lens.
  Other Names: ZCB00
  Arms: Monofocal Intraocular Lens

SUMMARY:
The purpose of this study is to evaluate near vision of the One-Piece Tecnis Multifocal lens (ZMB00) vs. the One-piece Tecnis monofocal lens (ZCB00)and additionally evaluate general postoperative outcomes of the One-Piece Tecnis Multifocal lens.

ELIGIBILITY:
Inclusion Criteria:

* bilateral cataracts and otherwise healthy eyes
* visual potential of Decimal 0.8 in each eye

Exclusion Criteria:

* any medications affecting vision
* any chronic disease/illness that would affect risk to subject or outcomes of the study
* any ocular pathology/abnormalities that may affect visual outcomes or confound study results
* desire for monovision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szurman, PD Dr. med., Principal Investigator

RESULTS

PARTICIPANT FLOW:
Groups:
- ZMB00 Multifocal Intraocular Lens: Subjects bilaterally implanted with the Model ZMB00 Multifocal Intraocular Lens
- ZCB00 Monofocal Intraocular Lens: Subjects bilaterally implanted with the Model ZCB00 Monofocal Intraocular Lens
Period: Overall Study
Arm/Group | ZMB00 Multifocal Intraocular Lens | ZCB00 Monofocal Intraocular Lens
Started | 36 | 34
Completed | 33 | 31
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Not implanted bilaterally | 2 | 1

BASELINE CHARACTERISTICS:
Population: A total of 34 ZMB00 multifocal and 33 ZCB00 monofocal subjects were implanted bilaterally. Data analysis for baseline characteristics was completed on these 67 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | ZMB00 Multifocal Intraocular Lens | ZCB00 Monofocal Intraocular Lens | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] — A total of 34 ZMB00 multifocal and 33 ZCB00 monofocal subjects were implanted bilaterally. Data analysis for baseline characteristics was completed on these 67 subjects.
  years | 63.1 (11.4) | 68.3 (11.3) | 65.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants] — A total of 34 ZMB00 multifocal and 33 ZCB00 monofocal subjects were implanted bilaterally. Data analysis for baseline characteristics was completed on these 67 subjects.
  Participants
    Female | 23 | 17 | 40
    Male | 11 | 16 | 27

OUTCOME MEASURES:

1. Secondary Outcome: Number of Subjects With 20/40 or Better Best Corrected Binocular Distance Visual Acuity
Time Frame: 4-6 months
Population: Within the 4-6 month time frame, one assessment was performed per participant. Though 70 subjects started the study (36 ZMB00; 34 ZCB00), best corrected binocular diatance visual acuity data were available for only 32 ZMB00 and 31 ZCB00 subjects at the the 4-6 month visit.
Measure: Number; unit: participants
Arm/Group | ZMB00 Multifocal Intraocular Lens | ZCB00 Monofocal Intraocular Lens
Number analyzed (Participants) | 32 | 31
participants | 32 | 31

2. Primary Outcome: Mean LogMAR Binocular Photopic Distance Corrected Near Visual Acuity at 33 cm
Description: Snellen equivalent for the mean logMAR binocular photopic distance corrected near visual acuity at 33 cm is 20/24 for the Multifocal Group. Snellen equivalent for the mean logMAR binocular photopic distance corrected near visual acuity at 33 cm is 20/81 for the Monofocal Group.
Time Frame: 4-6 Months
Population: Within the 4-6 month time frame, one assessment was performed per participant. Though 70 subjects started the study (36 ZMB00; 34 ZCB00), data for logMAR binocular photopic distance corrected near visual acuity at 33 were available for only 33 ZMB00 and 31 ZCB00 subjects at the the 4-6 month visit.
Measure: Mean (Standard Deviation); unit: logMAR visual acuity
Arm/Group | ZMB00 Multifocal Intraocular Lens | ZCB00 Monofocal Intraocular Lens
Number analyzed (Participants) | 33 | 31
logMAR visual acuity | 0.07 (0.12) | 0.61 (0.15)

ADVERSE EVENTS:
Arm/Group | ZMB00 Multifocal Intraocular Lens | ZCB00 Monofocal Intraocular Lens
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 3/36 | 4/34
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZMB00 Multifocal Intraocular Lens (N=36) | ZCB00 Monofocal Intraocular Lens (N=34)
Macular edema (Eye disorders) | 1 (1) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0)
IOL replacement secondary to broken haptic during surgery (Eye disorders) | 0 (0) | 1 (1)
Wound leakage (Eye disorders) | 0 (0) | 1 (1)
Head injury secondary to car accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head and shoulder injury secondary to wheelchair malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other